CLINICAL TRIAL: NCT05882851
Title: Investigation of the Effect of Nutrition and Risk Factors on the Failure of Vaginitis Treatment
Brief Title: Effect of Nutrition in the Treatment of Vaginitis
Status: Completed | Type: Observational
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, AYBALA TAZEOGLU, assistant professor, Osmaniye Korkut Ata University
Other Study IDs: OsmaniyeKAUnad
Record Dates: First submitted 2023-04-11; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Vaginitis
Keywords: vaginitis; carbohydrates; treatment; risk factors
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- grup 1: Those who recover after vaginitis treatment
  Interventions: Behavioral: determination of the current nutritional status of patients
- grup 2: those who were resistant to treatment
  Interventions: Behavioral: determination of the current nutritional status of patients

INTERVENTIONS:
Behavioral: determination of the current nutritional status of patients — No intervention was made on the patients. Nutritional status was recorded during the treatment process. Current nutritional status and other risk factors were compared according to recovery status after treatment.

SUMMARY:
Vaginitis is an inflammation or infection of the vagina. It is successfully treated for causative pathogenesis. However, it can be recurrent or treatment-resistant vaginitis. The investigator's aim in this study is to investigate the effect of nutrition and risk factors on the failure of vaginitis treatment.

DETAILED DESCRIPTION:
Predictively investigated patients diagnosed with vaginitis in the Gynecology and Obstetrics Clinic between January 2022 and April 2022. Patients with a diagnosis of vaginal infection, which were planned for medical treatment, who came for a follow-up examination, whose treatment effectiveness was re-evaluated, and whose data were complete were included in the study. Patients with co-existing gynecological diseases, who did not use the recommended medical treatment regularly, did not come to the follow-up examination within the recommended time, and could not evaluate the effectiveness of the treatment were excluded from the study.

The Obstetrician and Gynecologist gave medical treatment to all patients diagnosed with vaginal infection. The patient was called for control two weeks later. The patients included in the study were divided into two groups, those who recovered after treatment (group 1) and those who were resistant to treatment (group 2) and were compared.

Demographic data (age, gender), menopause, presence of diabetes mellitus, medical history, body mass index (BMI), total body fat and abdominal fat ratio, daily fiber consumption, carbohydrate percentage in the diet, and simple sugar ratio were recorded for the patients included in the study. In addition, the presence of birth in her medical history, delivery technique (vaginal, cesarean section), and history of recurrent vaginitis were questioned and recorded.

Anthropometric measurement Body weight and height measurements of the patients were made. Body mass index was calculated as weight (kilograms) / height squared (square meters).

Body fat measurement TANITA device is a device with 8 electrodes, working with 50 kHz constant current (hand to hand, foot to foot), measuring fat ratio, muscle mass and lean mass value for five different regions (right and left arm, right and left leg, trunk) with 5 different current waves. The measurements were carried out considering the working principles of the bioelectrical impedance analysis (BIA) device. Total body fat and abdominal fat ratio were measured with Tanita. Measurements were calculated as a percentage (%) and recorded.

Nutritional Consumption Record (BeBiS). In the study, information about the patient's diet and the carbohydrate, fat and protein ratios consumed in the diet was obtained by questioning the daily consumed foods when the patient came to the control. The three-day food consumption of the patients was recorded using the BeBis program. First, the percentage of carbohydrates and simple sugars (%) of dietary food intake was calculated and recorded. In addition, the daily pulp consumption amount (grams) was recorded.

ELIGIBILITY:
Inclusion criteria:

* admitted to the Gynecology and Obstetrics Clinic with a diagnosis of vaginal infection and medical treatment was planned,
* regular check-up
* agreeing to participate in the research,
* not pregnant
* over 18 years old

Exclusion Criteria:

* under 18 years old,
* pregnant,
* who refused to participate in the research,
* who did not come to their check-ups on time for treatment
* who did not come to their check-ups on time for treatment
* diagnosed with a psychiatric disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Vaginitis is a gynecological disease.
Study Population: Female patients over the age of 18 with a diagnosis of vaginal infection.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
determination of the current nutritional status of patients | up to 1 week
  Three-day food consumption of the patients was recorded using the BeBis program. First, daily consumption of carbohydrates, proteins, fats was recorded in grams, and the percentage of carbohydrates and simple sugars (%) of total energy intake was calculated and recorded. In addition, daily pulp consumption amount (gram) was recorded.

SECONDARY OUTCOMES:
comparison of vaginitis treatment results and nutritional analysis results, determination of the effect of nutrition on treatment | up to 3 week
  At the end of the four-week medical Vaginitis treatment administered by the doctor, the patients who responded positively to the treatment and were resistant to the treatment were divided into groups and the results of the food consumption analysis on Bebis were carbohydrate, protein, fat consumption amount (gram), the percentage of carbohydrate and sugar in total energy, and other risk factors (the presence of birth in The effects of macronutrients and simple sugar consumption on the treatment of vaginitis were determined by comparing each medical history, delivery technique (vaginal, cesarean section), and history of recurrent vaginitis were questioned and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Aybala Tazeoğlu, Merkez, Osmaniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want the plan to be known.

REFERENCES:
- [Background] Koumans EH, Sternberg M, Bruce C, McQuillan G, Kendrick J, Sutton M, Markowitz LE. The prevalence of bacterial vaginosis in the United States, 2001-2004; associations with symptoms, sexual behaviors, and reproductive health. Sex Transm Dis. 2007 Nov;34(11):864-9. doi: 10.1097/OLQ.0b013e318074e565. PMID 17621244
- [Background] Thoma ME, Klebanoff MA, Rovner AJ, Nansel TR, Neggers Y, Andrews WW, Schwebke JR. Bacterial vaginosis is associated with variation in dietary indices. J Nutr. 2011 Sep;141(9):1698-704. doi: 10.3945/jn.111.140541. Epub 2011 Jul 6. PMID 21734062
- [Background] Sheard NF, Clark NG, Brand-Miller JC, Franz MJ, Pi-Sunyer FX, Mayer-Davis E, Kulkarni K, Geil P. Dietary carbohydrate (amount and type) in the prevention and management of diabetes: a statement by the american diabetes association. Diabetes Care. 2004 Sep;27(9):2266-71. doi: 10.2337/diacare.27.9.2266. No abstract available. PMID 15333500
- [Background] Collins SL, McMillan A, Seney S, van der Veer C, Kort R, Sumarah MW, Reid G. Promising Prebiotic Candidate Established by Evaluation of Lactitol, Lactulose, Raffinose, and Oligofructose for Maintenance of a Lactobacillus-Dominated Vaginal Microbiota. Appl Environ Microbiol. 2018 Feb 14;84(5):e02200-17. doi: 10.1128/AEM.02200-17. Print 2018 Mar 1. PMID 29269494